CLINICAL TRIAL: NCT04274998
Title: Evaluation of in Vivo Neuroinflammation in Alzheimer's Disease Using Novel Positron Emission Tomography (PET/CT) Imaging
Brief Title: Neuroinflammation Imaging in AD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 834090
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Healthy Volunteer
MeSH Terms: conditions — Alzheimer Disease | interventions — Fluorine-18; (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AD/MCI or HC (Experimental): Main Study: Subjects are diagnosed with Alzheimer's Disease (AD)/Mild Cognitive Imparment (MCI) or are healthy volunteers/controls (HC).
  Interventions: Drug: [18F]NOS
- AD/MCI or HC with Genetic Polymorphism (Experimental): Sub-Study: Subjects have a specific genetic polymorphism andare diagnosed with Alzheimer's Disease (AD)/Mild Cognitive Imparment (MCI) or are healthy volunteers/controls (HC).
  Interventions: Drug: [11C]PBR28

INTERVENTIONS:
Drug: [18F]NOS — Main Study: PET/CT imaging will be used to evaluate neuroinflammation in the brain using the investigational radiotracer [18F]NOS.
  Arms: AD/MCI or HC
Drug: [11C]PBR28 — Sub-Study: Additional PET/CT imaging will be used to evaluate neuroinflammation in the brain for subjects with specific genetic polymorphism using the investigational radiotracer [11C]PBR28 in comparison to [18F]NOS.
  Arms: AD/MCI or HC with Genetic Polymorphism

SUMMARY:
This research study is being done to learn more about inflammation in the brain using Positron Emission Tomography/Computed Tomography (PET/CT) imaging in people with Alzheimer's Disease/Mild Cognitive Impairment or healthy controls.

If the subject agrees to be in this study, she/ he will have a PET/CT scan using the investigational radiotracer [18F]NOS. A subject with a specific genetic polymorphism may also agree to be in the sub-study in which she/he will have another PET/CT scan using the investigational tracer [11C]PBR28 for comparison with the FNOS [18F]NOS scan. For subjects who agree to this sub-study they may undergo the brain PET/CT scan with [11C]PBR28 either on the same day as the [18F]NOS PET/CT or on another day. The subject may have a screening visit before the PET/CT scan visit if the investigator needs to confirm the subject is able to be in the study.

A blood sample will be taken before the scans. Additional blood samples will be taken during the PET scans. Subjects must also agree to have an MRI scan for this research study if she/he has not had a recent scan that the study doctor decides can be used for this study.

ELIGIBILITY:
Inclusion Criteria (HC cohort only):

1. - Males and females ≥ 55 years of age
2. Part of the UPenn ADC research cohort with designation of cognitively normal per ADC database.
3. A brain amyloid PET scan ≤ 1 year prior to enrollment in this study that is determined to be negative by the study PI.
4. Mini-mental status exam (MMSE) score of 28 or higher per ADC database.
5. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Inclusion Criteria (AD/MCI cohort only)

1. Males and females ≥ 55 years of age
2. Part of the Upenn ADC research cohort with designation that the presence of Alzheimer's pathology is likely per ADC database.
3. A brain amyloid PET scan ≤ 1 year prior to enrollment in this study that is determined to be positive by the study PI.
4. Mini-mental status exam (MMSE) score of 14-27 per ADC database.
5. Subjects must have a designated study partner to accompany them to study visits

Inclusion Criteria 11C-PBR28 sub-study (both HC and AD/MCI cohorts)

1. High affinity carrier of the rs6971 TSPO polymorphism (whole genome sequencing is available from the UPenn ADC research cohort and will be interrogated for this polymorphism)

Exclusion Criteria (HC and PD cohorts):

1. Females of child-bearing potential will not be included, female subjects must be post-menopausal or surgically sterile
2. History of epilepsy or seizure disorder as assessed by medical record review and/or self-report
3. History of head trauma or evidence of structural abnormalities such as a major stroke or mass on MRI that in the opinion of an investigator may interfere with the uptake of applicable radiotracer as assessed by medical record review and/or self-report
4. Current tobacco or nicotine dependence. History of greater than 5 pack years of smoking and less than 2 years since smoking cessation.
5. Have a history of significant or ongoing alcohol abuse or substance abuse or dependence based on medical record review or self-reported
6. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
7. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician or investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Understanding the uptake of [18F]NOS in the human brain in AD/MCI and Healthy Controls | 3 years
  This main study outcome measure will be comparison of whole brain GM binding between controls and the MCI/AD group. the investigator will compare groups with a t-test. the investigator will evaluate the correlation of whole brain GM binding of 18F-NOS.
Comparing the patterns of [18F]NOS brain uptake with patterns of cerebral amyloidosis and neurodegeneration using PET/CT | 3 years
  This main study outcome measure will include regional and voxel-wise comparisons between binding of the tracers. Correlation between regional 18F-NOS binding and either amyloid PET SUVR (calculated with cerebellar gray matter reference) or GM volumetric measurements will be evaluated using Pearson's r and rank sum correlation initially using false discovery rate (FDR)-corrected<0.05 statistical thresholds

SECONDARY OUTCOMES:
Understanding the uptake of [11C]PBR28 in the human brain in AD/MCI and Healthy Controls with a specific genetic polymorphism | 3 years
  This sub-study outcome measure will be comparison of whole brain GM binding between controls and the MCI/AD group. the investigator will compare groups with a t-test. the investigator will evaluate the correlation of whole brain GM binding of 11C-PBR28
Comparing the patterns of [11C]PBR28 brain uptake with patterns of cerebral amyloidosis and neurodegeneration using PET/CT | 3 years
  This sub-study outcome measure will include regional and voxel-wise comparisons between binding of the tracers. Correlation between regional 11C-PBR28 binding and either amyloid PET SUVR (calculated with cerebellar gray matter reference) or GM volumetric measurements will be evaluated using Pearson's r and rank sum correlation initially using false discovery rate (FDR)-corrected<0.05 statistical thresholds

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States